CLINICAL TRIAL: NCT02641080
Title: Evaluating the Need for Pneumatic Compression Devices: A Randomized-controlled Trial (RCT) of Aspirin Versus Aspirin and Pneumatic Compression Devices
Brief Title: Evaluating the Need for Pneumatic Compression Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Matthew Dietz, MD, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1508807749
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Participants randomized to aspirin alone will be advised to take a 325mg per day as their outpatient DVT/PE prophylaxis.
  Interventions: Drug: Aspirin
- Aspirin with portable Compression Device (Active Comparator): Participants randomized to the compression device group are asked to wear the compression devices for 20 hours a day for 2 weeks along with taking an 325mg aspirin per day as their outpatient DVT/PE prophylaxis.
  Interventions: Drug: Aspirin; Device: Portable Compression Device

INTERVENTIONS:
Drug: Aspirin — If there is evidence that aspirin alone is equivocal to using both the pumps and aspirin, this could lower health care cost and burden for patients undergoing total joint arthroplasty while establishing that the rate of DVT/PE does not increase with the absence of the compression device.
  Other Names: ASA
Device: Portable Compression Device — If there is evidence that aspirin alone is equivocal to using both the pumps and aspirin, there could be lower health care cost and burden for patients undergoing total joint arthroplasty while establishing that the rate of DVT/PE does not increase with the absence of the compression device.
  Arms: Aspirin with portable Compression Device

SUMMARY:
For patients undergoing total hip and knee arthroplasty, does the use of Aspirin alone compared to using Aspirin along with a mobile compression device provide equivocal results for preventing Deep Vein Thrombosis (DVT) and pulmonary embolism (PE) after total joint arthroplasty? The investigator will evaluate the prevention of DVT/PE after total hip and knee arthroplasty will be evaluated to see if there is a decreased risk of bleeding while continuing to prevent thromboembolic disease. The equivalency of using the mobile compression devices with aspirin compared to aspirin alone in patients undergoing total hip and knee arthroplasty will be evaluated. A previous study has shown that patient compliance with the pneumatic compression device is less than 80%.

DETAILED DESCRIPTION:
The research question is: does the use of Aspirin alone compared to using Aspirin along with a mobile compression device provide equivocal results for preventing Deep Vein Thrombosis (DVT) and pulmonary embolism (PE) after total joint arthroplasty? Participants were randomized to either receive aspirin and mobile pneumatic compression devices or aspirin alone as outpatient DVT prophylaxis as their standard of care after primary total hip and total knee arthroplasty. Participants randomized to the compression device group were asked to wear the compression devices for 20 hours a day for 2 weeks along with taking an aspirin (325mg once a day), per standard of care. Participants randomized to aspirin alone took 325 mg per day. Participant usage information from Active Care +S.F.T. mobile devices was collected. The information was recorded at the participant's first follow up visit occurring between 7-21 days post-surgery. All of the participants were asked to keep a checklist indicating aspirin intake compliance each day, which was returned at their first follow up visit. Participants randomized to mobile pneumatic compression device and aspirin (325 mg) were asked to complete a satisfaction questionnaire about the compression device at their first follow up visit. Participants received a phone call from a member of the research team approximately 90 days post-op. The call was necessary to assess if any participants have been diagnosed with DVT at another hospital.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18+ years of age, scheduled at WVU Medicine Center for Joint Replacement for a History and Physical visit to undergo a total hip or knee surgery.
2. Primary replacements and revisions.
3. Weight bearing as tolerated postoperatively.

Exclusion Criteria:

1. History of DVT/PE
2. History of hypercoagulable disorder
3. Currently on other blood thinning medication with the exception of aspirin (Plavix, Coumadin, xarelto, pradaxa, lovenox, heparin, other Factor Xa inhibitors).
4. Patients less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Dietz, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Medicine Department of Orthopaedics, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin | Aspirin With Portable Compression Device
Started | 40 | 40
Completed | 38 | 33
Not Completed | 2 | 7
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Rehab Center denied use of pumps | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Aspirin With Portable Compression Device | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.0) | 60.8 (13.0) | 61.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 25 | 43
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 40 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 38 | 40 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
TKA/THA Enrollment [Count of Participants; unit: Participants]
  Total Knee | 19 | 22 | 41
  Total Hip | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolism
Description: Patients clinically diagnosed with a DVT or PE during the immediate 90 days post operative.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Aspirin With Portable Compression Device
Number analyzed (Participants) | 40 | 40
Participants | 0 | 3

2. Secondary Outcome: Aspirin Usage Over 6 Week Post op Period
Description: Number of Participants Taking aspirin over the 6 week post op period
Time Frame: 6 week post op
Measure: Number; unit: participants
Arm/Group | Aspirin | Aspirin With Portable Compression Device
Number analyzed (Participants) | 40 | 40
participants | 2 | 1

3. Secondary Outcome: Compression Pump Compliance Over 2 Weeks Post op
Description: Patients found to be compliant with recommended pump use over the course of two weeks. Compliance is defined as the recommended dose of 20 hours during the recommend course of prophylaxis.
Time Frame: 14 days post operative
Population: The outcome measure is specific only to those who used a compression device, the 'aspirin with portable compression device' group. The 'aspirin only group' did not use the compression device.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Aspirin With Portable Compression Device
Number analyzed (Participants) | 0 | 39
Participants |  | 10

4. Secondary Outcome: Overall Pump Experience After 2 Weeks
Description: Correlation of Recorded Pump Compliance with perceived Patient Factors
Time Frame: 2 weeks post op
Population: The outcome measure is specific only to those who used a compression device, the 'aspirin with portable compression device' group. The 'aspirin only group' did not use the compression device.
  The correlation between patient experience with pumps and average percent compliance.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Aspirin | Aspirin With Portable Compression Device
Number analyzed (Participants) | 0 | 40
correlation coefficient
  Overall Experience |  | 0.36 [0.01 to 0.63]
  Pumps were Noisy |  | 0.26 [-0.09 to 0.55]
  Pumps were Painful |  | 0.11 [-0.44 to 0.25]
  Pumps were Hot |  | -0.22 [-0.52 to 0.14]
  Pumps were Itchy |  | -0.25 [-0.55 to 0.11]
  Pumps were Difficult on/off |  | -0.12 [-0.46 to 0.24]
  Pumps were Tight |  | -0.23 [-0.53 to 0.13]
  Pumps caused Sweating |  | -0.1 [-0.44 to 0.26]
  Pumps caused Numbness |  | -0.23 [-0.53 to 0.13]
  Pumps caused Skin irritation |  | 0.12 [-0.23 to 0.45]
  Pumps caused Tripping/Falling |  | -0.21 [-0.5 to 0.15]
  Pumps caused Insomnia |  | -0.12 [-0.45 to 0.24]
  Pumps felt like a massage |  | 0.05 [-0.3 to 0.4]
  Pumps were difficult to use |  | 0.44 [0.1 to 0.68]
  Pumps were comfortable |  | -0.27 [-0.51 to 0.15]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 3 months.
Description: No adverse events occurred in any participant enrolled in the study.
Arm/Group | Aspirin | Aspirin With Portable Compression Device
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No